CLINICAL TRIAL: NCT01627314
Title: A Phase 2 Controlled Trial of a Single ProHema®-CB Unit (Ex Vivo Modulated Human Cord Blood) As Part of a Double Umbilical Cord Blood Transplant Following Myeloablative or Reduced Intensity Conditioning For Patients Age 15-65 Years With Hematologic Malignancies.
Brief Title: The PUMA Trial is a Trial of a Single ProHema Modulated-Cord Blood (CB) Unit as Part of a Double CB Transplant in Patients With Hematologic Malignancies.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FT1050-03
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ProHema-CB with MAC Preparative Regimen (Experimental): ProHema-CB and Wash-Only CB Unit with myeloablative conditioning regimen (MAC)
  Interventions: Biological: ProHema-CB
- ProHema-CB with RIC Preparative Regimen (Experimental): ProHema-CB and Wash-Only CB Unit with reduced intensity conditioning regimen (RIC)
  Interventions: Biological: ProHema-CB
- Control Arm with MAC Preparative Regimen (Placebo Comparator): Two Wash-Only CB Units (Untreated CB) with myeloablative conditioning regimen
  Interventions: Biological: Untreated CB
- Control Arm with RIC Preparative Regimen (Placebo Comparator): Two Wash-Only CB Units (Untreated CB) with reduced intensity conditioning regimen
  Interventions: Biological: Untreated CB

INTERVENTIONS:
Biological: ProHema-CB — Ex-vivo CXCR4 upregulated hematopoietic progenitor cells, cord blood
  Arms: ProHema-CB with MAC Preparative Regimen; ProHema-CB with RIC Preparative Regimen
Biological: Untreated CB — Cord Blood
  Arms: Control Arm with MAC Preparative Regimen; Control Arm with RIC Preparative Regimen

SUMMARY:
This study is an open-label randomized, prospectively and historically controlled trial of the safety and efficacy of a single ProHema-CB unit used as part of a double CB transplant following myeloablative or reduced intensity conditioning for subjects age 15-65 years with hematologic malignancies. A maximum of 60 eligible subjects will be enrolled and treated in the trial at approximately 10 centers within the U.S.

DETAILED DESCRIPTION:
All subjects will receive a myeloablative or reduced intensity conditioning regimen, after which they will receive 2 Human Leukocyte Antigen (HLA)-matched or partially matched umbilical cord blood (UCB) units. A total of 40 subjects will receive one ProHema-CB as part of a double CB transplant and an additional 20 subjects will be enrolled as concurrent controls. The determination of which CB unit will be the ProHema-CB unit will be made based primarily upon the degree of HLA match.

ELIGIBILITY:
Inclusion:

1. Patients with hematologic malignancies for whom allogeneic stem cell transplantation is deemed clinically appropriate. Eligible diseases and stages include:

   1. Acute lymphoblastic leukemia (ALL) (including T lymphoblastic lymphoma) in complete remission (CR).

      • Remission is defined as < 5% blasts with no morphological characteristics of acute leukemia in a bone marrow with > 5% cellularity.
   2. Myelodysplastic disease, International Prognostic Scoring System (IPSS) Intermediate-2 or High risk (e.g., refractory anemia with excess blasts (RAEB), refractory anemia with excess blasts in transformation (RAEBt) or refractory anemia with severe pancytopenia or high risk cytogenetics. Patients have to have received leukemia type induction chemotherapy within ≤ 3 months and with ≤ 10% blasts by a bone marrow aspirate; a single hypomethylating agent is not considered adequate cytotoxic chemotherapy; all subtypes except chronic myelomonocytic leukemia (CMML).
   3. Acute myelogenous leukemia (AML) in high risk first CR or second or subsequent CR.

      * High risk first CR is defined by but is not limited to at least one of the following factors: greater than one cycle of induction chemotherapy to achieve CR, prior myelodysplastic syndrome (MDS), presence of fms-like tyrosine kinase 3 (FLT3) abnormalities, French-American-British (FAB) M6 or M7 subtypes of leukemia, or adverse cytogenetics.
      * Remission is defined as < 5% blasts with no morphological characteristics of acute leukemia (e.g. Auer Rods) in a bone marrow with > 5% cellularity.
      * AML arising from myelofibrosis is not permitted.
   4. Biphenotypic/undifferentiated leukemia in first or subsequent CR (same definition of CR as for ALL/AML).
   5. Chronic myelogenous leukemia (CML) with prior exposure to cytotoxic chemotherapy for the treatment of blast phase or with demonstrated intolerance to at least 2 tyrosine kinase inhibitors.
   6. Non Hodgkin's lymphoma (T cell, large cell or mantle cell) or Hodgkin's lymphoma in second or subsequent CR or in partial remission (PR) with documented chemosensitivity. In addition, marginal zone lymphoma or follicular lymphoma that has progressed after ≥ 2 therapies (excluding single agent rituximab).

      * If the myeloablative conditioning regimen is selected, a history of prior myeloablative procedure is not allowed.
      * If the reduced intensity conditioning regimen is selected, and the subject has had a prior autologous transplant, it must have taken place > 3 months from anticipated Day 0 visit.
2. Lack of suitable 5 6/6 HLA matched related or (if institutional guidelines dictate) suitable 8/8 HLA A, B, C, DRß1 matched unrelated donor; or unrelated donor not available within appropriate timeframe.
3. Both cord blood units (CBUs) are qualified by Fate Therapeutics
4. Age 15 to 55 years (myeloablative regimen) or 15 to 65 years (reduced intensity regimen)
5. Body weight > 45 kg
6. Investigator selection of conditioning regimen (myeloablative or reduced intensity)
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2.
8. Signed Institutional Review Board (IRB) approved Informed Consent Form (ICF).

Exclusion:

1. History of prior allogeneic transplantation
2. Cardiac disease: symptomatic congestive heart failure or evidence of left ventricular dysfunction (Ejection fraction < 50%) as measured by gated radionuclide ventriculogram or echocardiogram; active angina pectoris, or uncontrolled hypertension; history of myocardial infarction with depressed ejection fraction.
3. Pulmonary disease: symptomatic chronic obstructive lung disease, symptomatic restrictive lung disease, or corrected diffusing capacity for carbon monoxide (DLCO) of < 50% of predicted, corrected for hemoglobin.
4. Renal disease: serum creatinine > 2.0 mg/dl and calculated creatinine clearance < 40 mL/min.
5. Hepatic disease: serum bilirubin > 2.0 mg/dl (except in the case of Gilbert's syndrome or ongoing hemolytic anemia), aspartate aminotransferase (SGOT) or alanine aminotransferase (SGPT) > 5 × upper limit of normal.
6. Neurologic disease: symptomatic leukoencephalopathy, active central nervous system (CNS) malignancy or other neuropsychiatric abnormalities believed to preclude transplantation.
7. HIV antibody.
8. Uncontrolled infection.
9. Pregnancy or breast feeding mother.
10. Inability to comply with the requirements for care after allogeneic stem cell transplantation.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-07; Primary Completion 2016-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Rate of early neutrophil engraftment using Myeloablative Conditioning | Neutrophil engraftment < 26 days
  To determine the rate of neutrophil engraftment after a single ProHema-CB unit is used as part of a double CB transplant following myeloablative conditioning for subjects with hematologic malignancies.
Rate of early neutrophil engraftment using Reduced Intensity Conditioning | Neutrophil engraftment < 21 days
  To determine the rate of neutrophil engraftment after a single ProHema-CB unit is used as part of a double CB transplant following reduced intensity conditioning for subjects with hematologic malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Storgard, M.D., Study Director — Fate Therapeutics
Locations (11):
- United States (11):
  - City of Hope, Duarte, California
  - Emory University-Winship Cancer Institute, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute- Hematopoietic Stem Cell Transplant Program, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health Sciences, Portland, Oregon